CLINICAL TRIAL: NCT05481385
Title: Single Oral Administration, Randomized, Open, Crossover and Bioequivalence Study of Ezetimibe Tablets Under Fasting Conditions in Healthy Subjects
Brief Title: Bioequivalence Study of Ezetimibe Tablets Under Fed Conditions in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22FWX-CZYZ-005-01
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Pharmacokinetics; Safety
Keywords: Ezetimibe

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test preparation (Experimental): Ezetimibe tablets: specification: 10mg; Package specification: 7 pieces / plate, 1 plate / box; Produced and provided by Changzhou Pharmaceutical Factory Co., Ltd.
  Interventions: Behavioral: Test Preparation-Reference preparation-Reference preparation
- Reference preparation (Active Comparator): Ezetimibe Tablets Ezetrol ®; Specification: 10mg, packaging specification: 10 pieces / plate, 1 plate / box; Licensee: MSD Pharma (Singapore) PTE. Ltd
  Interventions: Behavioral: Reference preparation-Reference preparation-Test Preparation; Behavioral: Reference preparation-Test Preparation-Reference preparation

INTERVENTIONS:
Behavioral: Reference preparation-Reference preparation-Test Preparation — Under fed conditions, subjects randomly divided into RRT group were given one tablet of reference preparation first, and then one tablet of reference preparation after cleaning period, and then one tablet of test preparation after cleaning period.
  Arms: Reference preparation
Behavioral: Reference preparation-Test Preparation-Reference preparation — Under fed conditions, subjects randomly divided into RTR group were given one tablet of reference preparation first, and then one tablet of test preparation after cleaning period, and then one tablet of reference preparation after cleaning period.
  Arms: Reference preparation
Behavioral: Test Preparation-Reference preparation-Reference preparation — Under fed conditions, subjects randomly divided into RTR group were given one tablet of test preparation first, and then one tablet of reference preparation after cleaning period, and then one tablet of reference preparation after cleaning period.
  Arms: Test preparation

SUMMARY:
The fed bioequivalence test adopts the experimental design of single center, single oral administration, random, open, two sequence, two cycle crossover and self-control.

DETAILED DESCRIPTION:
To investigate the in vivo pharmacokinetic characteristics of ezetimibe tablets (specification 10mg) in Chinese healthy subjects after a single oral administration under fed conditions, and to evaluate the bioequivalence of ezetimibe tablets produced by Changzhou Pharmaceutical Factory Co., Ltd. and the licensee MSD Pharma (Singapore) PTE. Ltd. To study the safety of single oral ezetimibe tablets (specification 10mg) in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male or female aged 18 and above.

  * The body mass index is in the range of 18.6-28.5 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
  * The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG, breath test for alcohol, drug abuse test.
  * The subjects have no family planning within 3 months and could select contraceptive method.
  * Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* • Being allergy to the study medications, smoking, alcohol abuse.

  * Participation in another clinical trial within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 96 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 96 hours
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 96 hours
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of abnormal blood pressure | 33 days
  Monitor both systolic and diastolic blood pressure
Incidence of abnormal temperature | 33 days
  Monitor the temperature
Incidence of abnormal pulse | 33 days
  Monitor the pulse
Incidence of abnormal electrocardiogram waveform | 33 days
  Electrocardiogram inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I clinical research center, Qingdao, Shandong, China